CLINICAL TRIAL: NCT06427759
Title: Optimizing Aesthetic Outcome for Arm Contouring Surgery by Utilizing Anthropometric Measurements
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abdelrahman Mostafa Shehata Mohammed (Other)
Responsible Party: Sponsor-Investigator, Abdelrahman Mostafa Shehata Mohammed, assistant lecturer, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 241094084
Record Dates: First submitted 2024-05-08; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Arm Aesthetics
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Intervention Model Description: Optimizing Aesthetic Outcome for Arm Contouring Surgery by Utilizing Anthropometric Measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anthropometric measures (No Intervention): *Group (A) Inclusion criteria of study: Anthropometric databases and studies done on females with normal BMI, In reproductive period , No history of pregnancy or weight fluctuation , No medical comorbidities .
- arm aesthetic surgery (Experimental): * Group (B) Include patients asking for arm aesthetic surgery .
  * Group B1: patients will be submitted for liposuction of arms only.
  * Group B2: patients will be submitted for liposuction and brachioplasty in same setting.
  * Group B3: patients will be submitted for liposuction then brachioplasty after 3 months.
  Interventions: Procedure: arm aesthetic surgery

INTERVENTIONS:
Procedure: arm aesthetic surgery — liposuction of arms brachioplasty of arms
  Other Names: liposuction, brachioplasty
  Arms: arm aesthetic surgery

SUMMARY:
Brachioplasty is a popular plastic surgery procedure. Current and common various techniques are based on either surgeon 's sense preoperatively. A method is needed to define how much skin and soft tissue should be excised precisely, or what can be a reference point to design a brachioplasty mathematically.(1)

Anthropometric reference measurements can be applied in designing arm aesthetic surgery.

Classically, anthropometry binds the upper arm length with forearm circumference and upper arm circumference to make postoperative results more harmonious and natural . (2)a 2020).

DETAILED DESCRIPTION:
2.4.1- Type of the study: 2.4. 2- Study Setting: Plastic and Reconstructive Surgery Department, Assuit University Hospital 2.4. 3- Study subjects:

a. Inclusion criteria:

* Group (A) this group will be available for measurements only with no interventions needed.
* Group (B) Include patients asking for arm aesthetic surgery .
* Group B1: patients will be submitted for liposuction only. liposuction is the preferred approach, particularly in young patients after massive weight loss.
* Group B2: patients will be submitted for liposuction and brachioplasty in same setting. When skin laxity is excessive, even in young patients, an extensive arm-long operation that extends across the axilla and onto the lateral chest is indicated.
* Group B3: patients will be submitted for liposuction then brachioplasty after 3 months.

in borderline cases to take chance for skin retraction .

c. Sample Size Calculation: sample size was calculated using g power program version 3.1.9.7 in order to detect anthropometric measures of arm and compare these measures with post operative cases, assumed effect size 0.8 based on clinical assumption (novel study) , α error 0.2 power 0.8 and allocation 1:1:1 the sample size will be 40 patients for each group. 2.4.4 -Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …): Group (A) will be subjected to these measures

*Arm length : Lateral length from acromion to lateral epicondyle Medial length from axilla to medial epicondyle

*Arm circumference : upper arm circumference Mid arm Lower arm

* Forearm circumference at widest point Arm assessed with elbow flexed at 90 degree and shoulder abducted at 90 degree. Group (B) will be subjected to
* Group B1: patients will be submitted for liposuction only.
* Group B2: patients will be submitted for liposuction and brachioplasty in the same setting.
* Group B3: patients will be submitted for liposuction then brachioplasty after 3, 6 and 12 months.

Pre-operative Assessment:

1. Patient history.
2. History of massive weight loss or any operation
3. Preoperative investigations
4. Informed consent.
5. Pre-operative photography. operative technique :- 1- most patients will take general anaesthesia . 2- then sterilization with betadine solution . 3 - pt positioned in supine position . 4- patient will be subjected according to its group to group(A): after injection of tumescent fluids - waiting 15 minutes - liposuction will be done circumferential in arm with cannula 4 .

group(B): after injection of tumescent fluids in the medial part of arm only(excised part ) - waiting 15 minute - then excision of medial part according to pinch test .

group (C): after injection of tumescent fluids all around _ waiting 15 minutes - liposuction will be done circumferential in arm with cannula 4 .

excision of the excessed part medially will be done after 3 months .

Patients will be subjected to arm measures before and after operation

* Arm length :

Lateral length from acromion to lateral epicondyle Medial length from axilla to medial epicondyle

*Arm circumference : upper arm circumference Mid arm Lower arm

* Forearm circumference at widest point Arm assessed with elbow flexed at 90 degree and shoulder abducted at 90 degree
* Pinch Test:
* Excess skin :
* Site of maximum redundancy:(Upper - Middle - Lower) arm
* Grade of Lipodystrophy:

Grade 1 :minimal fat with no ptosis Grade 2A :moderate fat with ptosis less than 5 cm Grade 2B : moderate to severe fat with ptosis 5- 10 cm Grade 3: extreme fat with ptosis more than 10 cm Grade 4 : mild to moderate fat with ptosis more than 10 cm. (3) Then comparing of post operative measurements after 3 , 6 and 12 months with the anthropometric measures of group (A) .

ELIGIBILITY:
Inclusion Criteria:

* group A : Anthropometric databases and studies done on females with normal BMI, In reproductive period , No history of pregnancy or weight fluctuation , No medical comorbidities .
* group B :Include patients asking for arm aesthetic surgery .

  * Group B1: patients will be submitted for liposuction only.
  * Group B2: patients will be submitted for liposuction and brachioplasty in same setting.
  * Group B3: patients will be submitted for liposuction then brachioplasty after 3 months.

Exclusion Criteria:

* 1) Males 2) Athletes 3) Current morbidities

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Group(A) anthropometric measures of arm length , arm circumference and forearm circumference . Group (B) compare postoperative measures of arm length , arm circumference and forearm circumference with anthropometric measures of Group A | 3 years
  Group(A) anthropometric measures of arm length , arm circumference and forearm circumference .
  Group (B) compare postoperative measures of arm length , arm circumference and forearm circumference with anthropometric measures of Group A

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No